CLINICAL TRIAL: NCT03033459
Title: Enhancing Breastfeeding Initiation, Exclusivity, and Duration: Effects of Prenatal Lactation-Focused Motivational Interviewing
Brief Title: Prenatal Lactation-Focused Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1605123038
Record Dates: First submitted 2017-01-18; First posted 2017-01-26 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Breast Feeding; Lactation Puerperal Increased; Infant Behavior; Maternal Behavior
Keywords: breast feeding; motivational interviewing
MeSH Terms: conditions — Breast Feeding; Galactorrhea; Infant Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): Participants assigned to the Motivational Interviewing condition will receive an approximately 45 (± 5) minute intervention provided by a female masters-level supervised psychologist with training in Motivational Interviewing.
  Interventions: Behavioral: Motivational Interviewing
- Psychoeducation Control (Active Comparator): Participants who have been randomly assigned to participate in the attention-control group session will receive approximately 45 (± 5) minutes of psychoeducation on typical developmental stages and infant feeding methods. The psychoeducation will be provided by a female masters-level supervised psychologist.
  Interventions: Behavioral: Psychoeducation Control

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing (MI) is a psychosocial intervention designed to help individuals increase readiness for behavior change by increasing intrinsic motivation and resolving ambivalence. MI founders MI conversations help clients change behavior through identifying and resolving discrepancies between goal behaviors and actual behaviors. Behavior change is promoted through the elicitation of "change talk," or client-verbalized arguments for change. In MI, change talk is elicited through two major components: the therapeutic relationship, or the embodiment of the "spirit" of MI, and technical skill.
  Arms: Motivational Interviewing
Behavioral: Psychoeducation Control — Psychoeducation on infant development, age 0-15 months, brief education on breastfeeding.
  Arms: Psychoeducation Control

SUMMARY:
Breastfeeding is good for the health of both mother and baby, but many women do not breastfeed, or do not breastfeed for as long as the participant would like. The purpose of this study is to compare two types of interventions on how each impacts breastfeeding. The interventions will be given during the third trimester of pregnancy, and the intervention is individual (i.e., one therapist and one participant). The first intervention is Motivational Interviewing, a type of counseling. The second intervention, or "control group," is education on how babies grow and develop. There general aims of this study are to compare women in the Motivational Interviewing group and control group on how the participants plan to feed the babies, how much the participants learn about and the participants opinions about breastfeeding, and how much the participants learn about how babies grow and develop. In addition, the groups will be compared as to whether the participants start breastfeeding, and how the participants are feeding the baby when the baby is one month old.

DETAILED DESCRIPTION:
1. Recruitment efforts will be made in the community via advertisements, online advertisements (e.g., Craigslist, Facebook), and in-person at various clinics and health fairs in the geographic area.
2. Prospective participants will contact the investigators via email or by calling the study phone number listed on the advertisements or verbally expressing interest in-person.
3. Once a participant indicates interest by contacting study personnel, a 5-minute screening interview will be conducted with the prospective participant using the screening questionnaire to ensure eligibility criteria are met. For those who do not qualify or agree to participate, the age and reason for non-qualification or declination to participate will be recorded; any other data will be destroyed by shredding or electronic shredding. For those who do qualify, name and contact information will be kept confidential and maintained in a locked room.
4. Participants will be asked to rate on a scale of -10 to +10 about the certainty that the participants will provide exclusive breastmilk to the babies for first six months. Responses from this item will be used as the covariate in the covariate adaptive randomization technique.
5. Eligible subjects will be invited to participate in the study, either in an exam room at West Virginia University's Family Medicine's clinic, participant's home, private room in the Quin Curtis Center for Psychological Services, or in another agreed-upon community location (e.g., church). The location of the study procedures is chosen by the participant.
6. At the start of this session, participants will be given an overview of the study, and the researcher will go over the consent form with the participant.
7. Following consent procedures, video-recording will begin, and all participants will complete the prenatal interview. After this interview, participants will complete five self-report measures, which include the Infant Feeding Knowledge Form, the Iowa Infant Feeding Attitudes Scale, Brief Breastfeeding Attitudes Questions, Perinatal Anxiety Screening Scale, and the Knowledge of Infant Development Inventory.
8. Intervention

   1. Participants assigned to the MI condition will receive an approximately 45 minute intervention provided a masters-level supervised psychologist with training in Motivational Interviewing.
   2. Participants who have been randomly assigned to participate in the attention-control group session will receive approximately 45 minutes of psychoeducation on typical developmental stages and infant feeding methods.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Female
3. Pregnant
4. At least 27 weeks pregnant
5. Able to read, write, speak, and understand English
6. Has access to a phone (either mobile or landline)
7. Lives within driving distance of Morgantown, WV, or is willing to travel to a location that is within driving distance to Morgantown, WV

Exclusion Criteria:

1. Multiple pregnancy
2. Within one week of due date
3. Has any of the following conditions:

   * Developmental or intellectual disability
   * Schizophrenia
   * Untreated, active tuberculosis
   * Human immunodeficiency virus (HIV)/Acquired immunodeficiency syndrome (AIDS)
   * Human T-cell lymphotropic virus type I or type II
   * History of lumpectomy or radiation to breast
4. Uses or is dependent upon any of the following substances (Moretti, Lee, & Ito, 2000):

   * Heroin
   * Cocaine
   * Methamphetamines
   * Marijuana
   * Phencyclidine (PCP)
   * Non-prescription opioids (e.g., morphine, oxycodone, hydrocodone)
5. Undergoing any of the following medications/treatments (American Academy of Pediatrics, 2001):

   * Antiretrovirals
   * Cancer chemotherapy (e.g., antimetabolites)
   * Radiation therapy
   * Acebutolol
   * Atenolol
   * Bromocriptine
   * Aspirin (salicylates)
   * Ergotamine
   * Lithium
   * Phenobarbital
   * Primidone
   * Sulfasalazine (salicylazosulfapyridine)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-09; Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Breastfeeding status at 1 month postpartum, participant self-report via telephone interview | 1 month

SECONDARY OUTCOMES:
Confidence (scale of 0-10) | 1 day
  Participant self-report of confidence in breastfeeding, scale of 0-10
Importance (scale of 0-10) | 1 day
  Participant self-report of importance of breastfeeding, scale of 0-10
Knowledge of breastfeeding-Breastfeeding Knowledge Questionnaire (survey) | 1 day
Attitudes towards breastfeeding- Iowa Infant Feeding Attitudes Scale (survey) | 1 day
Knowledge of infant development- Knowledge of Infant Development Inventory (survey) | 1 day
Intention to breastfeed Self-reported intention to breastfeed at prenatal time point | 1 day
Initiation Whether participant initiated breastfeeding, participant self-report via telephone interview | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W McNeil, PHD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request to the PI (Daniel McNeil, PhD) upon completion of the study, by emailing dmcneil@wvu.edu AND sehayes@mix.wvu.edu